CLINICAL TRIAL: NCT04892186
Title: Effects of Myo-inositol on the Menstrual Cycle, Hyperandrogenism, Chronic Inflammatory Process and Carbohydrate Metabolism in Women With Polycystic Ovary Syndrome
Brief Title: Effects of Myo-inositol in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 23458719.6.0000.0068
Record Dates: First submitted 2021-03-08; First posted 2021-05-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovary Syndrome; Resistance, Insulin; Glucose Intolerance
Keywords: myo-inositol; metformin; polycystic ovary syndrome; resistance insulin; glucose intolerance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Glucose Intolerance | interventions — Inositol; Metformin

STUDY DESIGN:
Intervention Model Description: Comparative and non-inferiority study of myo-inositol in relation to metformin. They will be divided into two groups of 30 patients: Group I (control) - they will receive metformin, orally, three times a day; Group II (experiment) - they will receive myo-inositol 2g, orally, twice a day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myo-inositol (Experimental): 30 women with resistance insulin or glucose intolerance will receive myo-inositol 2g + folic acid 200mcg, orally, twice a day for 6 months.
  Interventions: Drug: Myo-inositol
- Metformin (Active Comparator): 30 women with resistance insulin or glucose intolerance will receive metformin 850 mg, orally, twice a day for 6 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Myo-inositol — 30 women with polycystic ovary syndrome and insulin resistance or glucose intolerance will used myo-inositol 2g + folic acid 200mcg twice daily for 6 months, having a re-evaluation every 3 months.
  Evaluation will be made by transvaginal ultrasound, abdominal ultrasound, inflammatory tests, hormonal tests, glycemic curve with insulin curve, lipid profile, body mass index, evaluation of abdominal and hip circumference.
  Arms: Myo-inositol
Drug: Metformin — 30 women with polycystic ovary syndrome and insulin resistance or glucose intolerance will used metformin 850 mg twice a day for 6 months, having a re-evaluation every 3 months.
  Evaluation will be made by transvaginal ultrasound, abdominal ultrasound, inflammatory tests, hormonal tests, glycemic curve with insulin curve, lipid profile, body mass index, evaluation of abdominal and hip circumference.
  Arms: Metformin

SUMMARY:
The study will be carried out at the hospital of the medical school of sao paulo (HC-FMUSP) and the goal is to compare the effects of the administration of myo-inositol in relation to the effects of metformin in women with Polycystic Ovary Syndrome and insulin resistance or glucose intolerance. Menstrual cycle, hyperandrogenism, chronic inflammatory process, carbohydrate metabolism, hepatic steatosis will be evaluated. In total, 60 women in the reproductive period, with a variable age between 18 and 36 years old will be recruited and randomized in two groups: intervention- myo-inositol for 6 months, control group will use metformin also for 6 months.

DETAILED DESCRIPTION:
The study will involve 60 women in the reproductive period, with a variable between 19 and 36 years old and diagnosed with polycystic ovary syndrome (PCOS), according to Rotterdam- European Society of Human Reproduction and Embryology (ESHRE) / American Society for Reproductive Medicine (ASRM) criteria defined in 2003 and revised in 2018, and insulin resistance (presence acanthosis nigricans) or glucose intolerance (fasting glycemia, glycated hemoglobin or 75g glycemic overload and blood glucose assessment after 2 hours). It is a comparative and non-inferiority study of myo-inositol in relation to metformin. They will be divided into two groups of 30 patients: Group I (control) - they will receive metformin 850 mg, orally, twice a day; Group II (experiment) - they will receive myo-inositol 2g + folic acid 200mcg, orally, twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 19 to 36 with diagnosis of PCOS and insulin resistance or glucose intolerance.

Exclusion Criteria:

* Previous use of any hormonal treatment in the past three months;
* Other causes of anovulation;
* Gynecological or other associated conditions (endometriosis, adenomyosis or diabetes mellitus);
* FSH (Follicle Stimulating Hormone) > 15 Ul / L (2nd to 5th day of the cycle);
* Beta-hcG (human chorionic gonadotropin) positive (pregnancy).

Ages: 19 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Menstrual cycle | 6 months
  Analysis of period calendar.
Change in glucose metabolism | Every 3 months for up to 6 months
  Glucose tolerance curve with insulin curve will be performed every 3 months.
Change in glycated hemoglobin | Every 3 months for up to 6 months
  Glycated hemoglobin will be performed every 3 months.
Change in ultrasound of the ovaries | 6 months
  Transvaginal ultrasound to assess ovarian volume (measured in cubic centimeters) will be done before and after treatment.
Change in antral follicle count | 6 months
  Ultrasound of the ovaries will be done before and after treatment for antral follicle count (all follicles from 2 to 9 mm will be measured)
Change in body mass index | Every 3 months for up to 6 months
  Body mass index (kg/m2) will be assessed every 3 months.
Change in Abdominal Circumference and Hip Circumference | Every 3 months for up to 6 months
  Abdominal circumference and hip circumference (measured in centimeters) will be assessed every 3 months.
Change in body weight in kilograms | Every 3 months for up to 6 months
  Patients will be weighed every 3 months (measured in kilograms).

SECONDARY OUTCOMES:
Assess adherence to treatment. | Every 3 months for up to 6 months
  Medication use diary will be delivered and will be reviewed every 3 months to assess adherence to treatment (good adherence will be considered use of more than 80% of the medication provided).
Side effects | Every 3 months for up to 6 months
  Questionnaire will be carried out every 3 months for patient to describe the 3 main side effects and how much they have hindered the treatment or not.
Hepatic steatosis | 6 months
  Initial liver ultrasound will be done and repeated after 6 months of treatment to assess the presence or absence of hepatic steatosis and classify it as mild (grade 1), moderate (grade 2) and severe (grade 3).
Liver enzymes | 6 months
  Liver enzymes (aspartate aminotransferase, alanine aminotransferase,alkaline phosphatase) will be collected before and after treatment
Chronic inflammatory process | 6 months
  Chronic inflammatory markers will be accessed by analyzing RNA messenger from cervical-vaginal cytology before and after treatment.
C-reactive protein | 6 months
  Chronic inflammatory process will be also evaluated by serum measurement of c-reactive protein before and after treatment.
Homocysteine | 6 months
  Serum homocysteine dosage will be done before and after treatment to help assess a chronic inflammatory process.
Change in Lipid Profile | Every 3 months for up to 6 months
  Serum dosage of the lipid profile (high density lipoprotein - HDL, low density lipoprotein - LDL , very low density lipoprotein - VLDL, triglycerides, total cholesterol) will be done every 3 months
Modified Ferriman-Gallwey Score | 6 months
  Modified Ferriman-Gallwey Score will be performed before and after treatment and patients with a score above 7 will be considered hirsute.
Hormonal dosage (FSH, LH, progesterone, estradiol) | 6 months
  Hormonal dosage (FSH - Follicle-stimulating hormone, LH - luteinizing hormone, progesterone, estradiol) will be preformed before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Chada Baracat, Phd, Principal Investigator — research coordinator
Locations (2):
- Brazil (2):
  - Hospital Das Clinicas - Fmusp, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No